CLINICAL TRIAL: NCT00316381
Title: Myocardial REGeneration by Intracoronary Infusion of Selected Population of stEm Cells in Acute Myocardial iNfarcTion. Randomized Multicenter Trial
Brief Title: Stem Cell Therapy to Improve Myocardial Function in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silesian School of Medicine (Other)
Collaborators: Ministry of Science and Higher Education, Poland (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REGENT; Grant PBZ-KBN-099/P05/2003
Record Dates: First submitted 2006-04-18; First posted 2006-04-20 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Myocardial Infarction
Keywords: stem cells; acute myocardial infarction; regeneration; left ventricular ejection fraction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Autologous bone marrow-derived stem cells

SUMMARY:
The purpose of the study is to compare the efficiency of a sorted subpopulation of CD34+/CXCR4+ cells and unselected bone marrow-derived progenitor cells in the treatment of patients with acute myocardial infarction and a low left ventricular ejection fraction.

DETAILED DESCRIPTION:
Aim is to compare the efficiency of sorted subpopulation of CD34+/CXCR4+ cells and unselected bone-marrow-derived progenitor cells in treatment of patients with acute myocardial infarction and low left ventricular ejection fraction. The subpopulation of CD34+/CXCR4+ cells most likely contains the tissue-specific stem cells likely to be involved in myocardial salvage/regeneration after ischemic injury. This approach is novel and original, because so far no study identified the type of cells that actually contribute to stem cell-induced improvement in myocardial function in patients with AMI which were treated with unselected population of cells. The REGENT trial (prospective, randomized, multicentre trial comparing unselected BM mononuclear cells and sorted CD34/CXCR4+ cells in patients with myocardial infarction and low left ventricular ejection fraction) successfully treated with primary percutaneous coronary angioplasty within 12 hours after the onset of chest pain. The cells are delivered by intracoronary infusion. Efficiency is assessed by cardiac magnetic resonance imaging, echocardiography and left ventricular angiography.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction treated successfully with primary coronary angioplasty
* Left ventricular ejection fraction less than 40%
* Informed consent granted

Exclusion Criteria:

* Presence of significant coronary stenoses in non-infarct related artery requiring revascularization
* Cardiogenic shock
* Previous myocardial infarction
* Age < 18 years and > 75 years
* Pregnancy
* Neoplasm
* Contraindications for MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction and volumes measured by echocardiography | 6 months
Left ventricular ejection fraction and volumes measured by angiography | 6 months

SECONDARY OUTCOMES:
Safety | 6, 12 months
Left ventricular function in dobutamine stress test | 6 months
Coronary flow reserve by adenosine MRI test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michal Tendera, MD, PhD, Principal Investigator — Third Division of Cardiology Silesian School of Medicine
Locations (4):
- Poland (4):
  - III Division of Cardiology Silesian School of Medicine, Katowice
  - Jagiellonian University Institute of Cardiology, Krakow
  - Poznan University of Medical Sciences II Clinic of Cardiology, Poznan
  - National Institute of Cardiology, Warsaw

REFERENCES:
- [Background] Wojakowski W, Tendera M, Michalowska A, Majka M, Kucia M, Maslankiewicz K, Wyderka R, Ochala A, Ratajczak MZ. Mobilization of CD34/CXCR4+, CD34/CD117+, c-met+ stem cells, and mononuclear cells expressing early cardiac, muscle, and endothelial markers into peripheral blood in patients with acute myocardial infarction. Circulation. 2004 Nov 16;110(20):3213-20. doi: 10.1161/01.CIR.0000147609.39780.02. Epub 2004 Nov 8. PMID 15533859
- [Background] Wojakowski W, Tendera M, Zebzda A, Michalowska A, Majka M, Kucia M, Maslankiewicz K, Wyderka R, Krol M, Ochala A, Kozakiewicz K, Ratajczak MZ. Mobilization of CD34(+), CD117(+), CXCR4(+), c-met(+) stem cells is correlated with left ventricular ejection fraction and plasma NT-proBNP levels in patients with acute myocardial infarction. Eur Heart J. 2006 Feb;27(3):283-9. doi: 10.1093/eurheartj/ehi628. Epub 2005 Nov 2. PMID 16267071
- [Background] Kucia M, Ratajczak J, Ratajczak MZ. Bone marrow as a source of circulating CXCR4+ tissue-committed stem cells. Biol Cell. 2005 Feb;97(2):133-46. doi: 10.1042/BC20040069. PMID 15656779
- [Derived] Dabrowski W, Tekieli L, Mazurek A, Lanocha M, Banys RP, Zmudka K, Majka M, Wojakowski W, Tendera M, Musialek P. Transcoronary stem cell transfer and evolution of infarct-related artery atherosclerosis: evaluation with conventional and novel imaging techniques including Quantitative Virtual Histology (qVH). Postepy Kardiol Interwencyjnej. 2022 Dec;18(4):483-495. doi: 10.5114/aic.2023.125609. Epub 2023 Feb 6. PMID 36967840